CLINICAL TRIAL: NCT03883295
Title: Evaluation of Clinical and Radiological Success of Vital Amputation Treatment Applied in Teeth With Irreversible Pulpitis Using MTA
Brief Title: Evaluation of Clinical and Radiological Success of Vital Amputation Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, ELİF KALYONCUOĞLU, Assoc.Prof, Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 352
Record Dates: First submitted 2019-03-18; First posted 2019-03-20 (Actual); Last update posted 2019-03-25 (Actual); Status verified 2019-03

CONDITIONS: Endodontic Inflammation; Pulp Disease, Dental
MeSH Terms: conditions — Pulpitis; Dental Pulp Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Experimental): root canal treatment will be initiated
  Interventions: Procedure: Control
- NeoMTA Plus (Experimental): vital pulp treatment using neomta plus will be used.
  Interventions: Procedure: NeoMTA Plus

INTERVENTIONS:
Procedure: Control — The specimens will be root canal treated conventionally
  Other Names: Conventional root canal treatment
  Arms: Control
Procedure: NeoMTA Plus — The specimens will be subjected to vital pulp amputation using NeoMTA Plus.
  Other Names: Pulp amputation
  Arms: NeoMTA Plus

SUMMARY:
Total amputation therapy; is a treatment method aimed at maintaining the vitality of the radicular pulp remaining as a result of complete removal of coronal pulp tissue. In cases where pulp is exposed due to caries or trauma, the pulp is vital, bleeding can be controlled during the procedure, no periapical pathology is seen and radicular pulp is healthy.

Traditionally, acute pulp pain is thought to be a symptom of irreversible pulpitis, and it is thought that there is little chance of the pulp returning to its normal situation after removal of the irritants. Root canal treatment has been accepted as the gold standard for the treatment of these symptoms. In recent studies, spontaneous or severe pain before procedure has not always indicated that pulp has no repair capacity, and deep carious lesions are not necessarily associated with irreversible pulpal pathology. Histological studies showed that even when caries reach the pulp or degeneration and inflammation were seen in it, there was a healthy section still present in the pulp. Therefore, it is stated that the healthy pulp remaining as a result of total amputation performed by removal of degenerated pulp can be preserved. Furthermore, it is stated that for the healing potential of the remaining pulp tissue, the original signal should be that the bleeding can be controlled after the amputation of the infected pulp tissue.

While the most popular method in the treatment of vital pulp is CaOH, the American Academy of Pediatric Dentistry has been reported to be more resistant to dissolution in the protocol in recent years. MTA is a more suitable material because it is more homogeneous, and forms a thicker dentin bridge. However, the MTA requires a long time to harden, it is difficult to manipulate and color. In recent years, researchers have focused on creating new MTA formulations to improve their physicochemical properties without affecting their biocompatibility and bioactivity.

NeoMTA Plus is a new fine powder tricalcium silicate. It consists of a water-based gel and powder mixture and the powder-gel mixing ratio may vary depending on the area of use. It is a material similar to MTA Plus. However, in order to avoid tooth discoloration, tantalium oxide used instead of the bismuth oxide and required calcium hydroxide used to induce the formation of mineralized tissue.

DETAILED DESCRIPTION:
This study was approved by the Ondokuz Mayis University Clinical Research Ethics Committee (OMU KAEK 2018/352) All clinical treatments will be carried out by two researchers as pediatricians for patients aged 8-18 years and endodontics specialists for patients over 18 years of age. All patients who have participated in the study will be informed by written and verbal information. In the study, two groups will be formed according to the two age groups. According to the results of power analysis, 95% confidence and 94.3% test power for each group 30 cases, in total 60 cases will be taken. Patients included in the study will be treated for lower molar and lower / upper premolar teeth. Five patients who underwent root canal treatment from each age group will be used as a control group to evaluate the dimensional changes of the root canal by the evaluation of their periapical radiograph.

The patient's age, gender, type of tooth, location and complaint of the patient will be recorded prior to clinical procedures. After clinical examination including percussion test, palpation test, vitality control, and periodontal examination, the radiographic evaluation will be completed by taking the periapical radiograph of the relevant tooth in parallel technique.

A local anesthetic solution containing 2% articaine hydrochloride (Ultraca from Sanofi Aventis, Istanbul, Turkey) will be applied to the tooth which will include, followed by isolation the tooth with rubber dam will be performed. Following the disinfection of the isolated tooth crown with 2% chlorhexidine gluconate, the current caries lesion will be removed under water cooling with the aid of sterile diamond drills and low-speed single-use steel rod drills, the teeth where the infected pulp has been completely removed but the pulp is not mechanically exposed. Indirect pulp treatment will be applied.

In case that the pulp is exposed while infected dentin is removed, the working protocol will be applied to the teeth. Accordingly, first, remove the dentin around the exposure area and remove the roof of the pulp chamber, then by using thick diamond drills under water cooling the coronal pulp until the level of the canal orifices will remove. To ensure hemostasis, sterile cotton pellets impregnated with 2.5% NaOCl will be kept 5min at the orifices of the canal. The procedure shall be repeated for a maximum of 3 times with a bleeding control every 5 minutes. At the end of 15 minutes, root canal treatment will be applied to the teeth where hemostasis is not provided. 2mm calcium silicate-based material (NeoMTA Plus) (Avalon Biomed Inc., Bradenton, FL, USA) will be placed on the expansive pulp tissue in the canal opening. In accordance with the manufacturer's instructions, NeoMTA Plus will be prepared by mixing a scale of powder with 1 drop of gel for 30 seconds and after being transported to the cavity, it will be lightly pressed with a damp cotton pellet and adapted to the base of the pulp chamber. The chemically curing glass ionomer will be applied as a cement base material. The enamel surfaces of the teeth will then be acidified for 30 seconds with 37% phosphoric acid for selective acidification. After the cavity is washed with plenty of water and dried at the humidity level, the binding agent (Single Bond Universal 3M / ESPE, USA) will be light-cured by applying to the enamel and dentin surface in 2 coats according to the company instructions. A nanoparticle composite (Filtek Ultimate, 3M / ESPE) will be applied to the cavity with 2 mm each layer technique and will be polymerized with the same LED device (Elipar FreeLight, 3M ESPE, Seefeld, Germany) for the 20s each layer. Following finishing and polishing operations, it will rebond the cavity limits. After the procedure, periapical radiograph will be taken again with parallel technique by using a film holder to ensure standardization from all teeth. All patients will be called up for follow-up every 3 months during the first year and then every 6 months. In the control, the relevant teeth shall be subjected to a cold test and an electrical pulp test (on the appropriate teeth). Also; the presence of postoperative pain, how long it will last, presence/absence of clinical symptoms, filling quality, presence of pulp obliteration will be evaluated. In addition, periapical radiograph will be taken with parallel technique. Assessments will be made by 2 researchers. Cohen kappa analysis will be conducted to evaluate the consistency between the researchers.

In situations where both clinical and radiographic findings are within normal limits will be recorded successfully. Pain, swelling, presence of sinus tract and presence of radiolucency in the periapical region will be recorded as a failure.

Radiographs taken from the patient by parallel technique will be recorded in digital environment and dimensional changes in root length, increase in dentin amount, the space of the root canal will be evaluated using Image J software program.

Statistical evaluation:

Statistical analysis of the data to be obtained:

The McNemar test was used for the statistical evaluation of the success levels for the time-dependent group. In the purpose of evaluation McNemar test , Two-Rate Z test will be applied to determine the differences between the groups (p <0.05).

ELIGIBILITY:
Inclusion Criteria:

* Having a lower molar and lower/upper premolars diagnosed with irreversible pulpitis

Exclusion Criteria:

* Patients with systemic disease
* Negative outcome of pulp sensibility
* Patients presenting abscess

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 70 (Estimated)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-12-15 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain | 12 months
  Using visual analogue scale by participant. It is usually presented as a 100-mm horizontal line on which the patient's pain intensity is represented by a point between the extremes of "no pain at all" and "worst pain imaginable". The scale has no other subscales.
Pulp sensibility | 12 months
  Using cold and electric pulp testings by clinicians
Radiological evaluation | 12 months
  Standardized periapical radiographs will be taken and monitored

CONTACTS AND LOCATIONS:
Overall Officials: Ayça T Ulusoy Yamak, Principal Investigator — ONDOKUZ MAYIS UNIVERSITY, FACULTY OF DENTISTRY DEPARTMENT OF PEDIATRIC DENTISTRY
Locations (1):
- Elif Kalyoncuoğlu, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No